CLINICAL TRIAL: NCT00712998
Title: Effect of X-Ray Computed Tomography Examination on the Blood Reactive Oxygen Species Level in Apparently Healthy Adults
Brief Title: X-Ray Computed Tomography and Blood Reactive Oxygen Species Level
Status: Terminated | Type: Observational
Why Stopped: Beacuse of unexpected administrative barriers, only 5 cases were enrolled in a year.
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Zei-Shung Huang, associate professor, Department of Internal Medicine, NTUH, National Taiwan University Hospital
Other Study IDs: 200803085R
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2008-03

CONDITIONS: Healthy
Keywords: radiation injuries; free radicals; reactive oxygen species; radiation injury from X-ray computed tomography; free radical production; blood reactive oxygen species level
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — only peripheral blood will be collected for measurement of reactive oxygen species.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Twenty subjects receiving health check program without X-ray computed tomography examination will be included as the control group.
- 2: Twenty subjects receiving health check program including X-ray computed tomography examination of lung will be included as the treatment group-1.
- 3: Twenty subjects receiving health check program including X-ray computed tomography examination of heart will be included as the treatment group-2.

SUMMARY:
The clinically widely used X-ray computed tomography examination has a low-grade radiation effect and recently has attracted much attention concerning the possible adverse effects of radiation on human body [ref. 1-5]. The radiation is harmful to human tissues and cells mainly because it can interact with water (which makes up to 80% of cells) to generate reactive oxygen species (ROS), especially the formation of hydroxyl radicals. So far as we can reach, there is no report concerning the relation between X-ray computed tomography examination and the blood ROS concentration. Therefore, we wish to conduct this study to clarify if the routinely applied X-ray computed tomography examination may induce a higher concentration of ROS in the peripheral blood.

Study subjects will be participants of health check program at our hospital. The only enrollment condition will be a scheduled X-ray computed tomography examination for either lung (20 cases) or heart (20 cases) of the study subject. Another 20 participants receiving health check program without X-ray computed tomography examination will be included as the control group. The formal consent will be delivered to the participants of health check program several days before their admission for health check and will be retrieved before the proceeding of health check.

Measurements and comparison of ROS concentration will be performed in the sampled peripheral blood before and after the performance of X-ray computed tomography examination during a regular health check program. Totally 120 blood samples will be collected from included 60 study subjects within 3 months. Reactive oxygen species（ROS）levels will be measured by a chemiluminescence (CL) analysing system (CLD-110, Tohoku Electronic Industrial, Sendai, Japan).

ELIGIBILITY:
Inclusion Criteria:

* Participants of health check program at our hospital who will receive a scheduled X-ray computed tomography examination for either lung (20 cases) or heart (20 cases).

Exclusion Criteria:

* Those whose age are under 50 or above 70 year-olds will be excluded.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participants of health check program at our hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-07 (Estimated); Study Completion 2008-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Zei-Shung Huang, MD, PhD, Principal Investigator — NTUH
Locations (1):
- NTUH, Taipei, Taiwan